CLINICAL TRIAL: NCT05985122
Title: Towards the Most Accurate Diagnosis and Monitoring of Complement-mediated Rare Kidney Diseases
Brief Title: New Analytic Tools for aHUS and C3G Diagnosis
Acronym: COMPRare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPRare-IRFMN
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hemolytic-Uremic Syndrome; Membranoproliferative Glomerulonephritis; Healthy
Keywords: Complement-mediated kidney diseases; Blood and tissue biomarkers; Assay standardization; Glycocalyx; Characterization of variants of unknown significance
MeSH Terms: conditions — Hemolytic-Uremic Syndrome; Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Intervention Model Description: The samples (healthy volunteers and HUS or MPGN patients) for the study will be identified between those of patients and healthy controls who provided consent to store their samples in the certified biobank of "Centro Daccò" (Centro di Risorse Biologiche Mario Negri - Biobanca Malattie Rare e Renali) for two previousely approved studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Patients diagnosed with C3G (15 positive and 15 negative for C3NEF) at Centro Daccò, will be identified between those who provided consent to store their samples in the certified biobank (UNI EN ISO 9001:2015; certification n° 6121) of "Centro Daccò" (Centro di Risorse Biologiche Mario Negri - Biobanca Malattie Rare e Renali) and to share them with external laboratories.
  Interventions: Diagnostic Test: C3NEF assay
- Healthy controls (Active Comparator): Healthy donors will be identified between those who provided consent to store their samples in the certified biobank (UNI EN ISO 9001:2015; certification n° 6121) of "Centro Daccò" (Centro di Risorse Biologiche Mario Negri - Biobanca Malattie Rare e Renali). Subject that meet the inclusion/exclusion criteria and for which there is no enough material stored in our biobank, will be recontacted by the investigators of "Centro Daccò" and, if agree, will be asked for serum sampling after informed consent signature.
  Interventions: Diagnostic Test: C3NEF assay

INTERVENTIONS:
Diagnostic Test: C3NEF assay — This assay will consist of a dual test, detecting C3 convertase binding C3NEF autoantibodies and measuring the functional consequence by complement alternative pathway (AP) activity using two distinct ELISA designs: C3NEF detection assay and AP activity assay.

SUMMARY:
This protocol is part of a larger project, COMPRare (COMPlement-mediated Rare kidney diseases), which has been financed on behalf of the EJP RD (European Joint Programme on Rare Diseases) program of EU and is leaded by a scientific consortium from 7 European countries.

The partners (P) of the consortium are:

P1. Radboudumc Amalia Children's Hospital (The Netherlands) P2. Semmelweis University (Hungary) P3. Cordeliers Research Center (France) P4. Max Delbruck Center for Molecular Medicine (Germany) P5. Istituto di Ricerche Farmacologiche Mario Negri (Italy) P6. Lund University (Sweden) P7. Lille University (France)

The general aim of the project is to define new diagnostic tools for complement activation in order to improve patients stratification and follow-up, thereby affecting time and choice of treatment in patients with aHUS and C3G.

Particularly, the specific objectives of the COMPRare are:

* To develop new standardized analytic assays thereby identifying specific complement prognostic biomarkers for early diagnosis, classification, improved monitoring and treatment of patients with aHUS and C3G;
* To in-depth characterize patients' complement abnormalities in blood, in patient-derived cells and in kidney biopsies;
* To identify strategies to classify VUS/LPV
* To find new pathophysiological pathways involved in aHUS and C3G for further improving disease diagnosis, monitoring and treatment.

The results of these studies will form the basis of personalized treatment with existing and upcoming complement inhibitory drugs for these rare complement-mediated kidney diseases.

DETAILED DESCRIPTION:
Atypical Hemolytic Uremic Syndrome (aHUS) and C3 Glomerulopathies (C3G) are ultra-rare conditions in which an uncontrolled complement activation results in renal inflammation with thrombotic microangiopathy (TMA) in aHUS and extensive deposition of complement fragments in the kidneys in C3G. In both conditions, these alterations lead to acute and chronic kidney damage and, ultimately, end-stage renal failure. The prevalence of genetic and acquired complement abnormalities varies between the two diseases, but covers mostly the same complement proteins. Blocking the complement system is the treatment of choice in aHUS and may have considerable potential in C3G, as evident from the increasing number of phase 3 trials with complement inhibitory drugs. Timely and accurate diagnosis is still challenging for clinicians, both for aHUS, to differentiate it from other forms of TMA, and for C3G, to distinguish it from other forms of glomerulonephritis (GN). In C3G, kidney biopsy is the diagnostic gold standard but it is not sufficient. Therefore, for both aHUS and C3G, there is an unmet need for accurate testing of genetic and acquired complement abnormalities. Moreover, interlaboratory complement-assays, in particular the tests for the C3 Nephritic Factors (C3NeFs; heterogeneous autoantibodies that stabilize the C3 convertase), vary considerably and, consequently, their standardization is a great necessity. Furthermore, the interpretation of genetic results in aHUS and C3G is not always conclusive.

Variants of Unknown Significance (VUS)/Likely Pathogenic Variant (LPV) in complement genes are often found in aHUS and C3G and require further characterization. A rapid and functional VUS/LPV determination and interpretation could help to better understand the disease pathophysiology and might influence diagnosis and treatment options.

Currently, aHUS patients are effectively treated with the complement C5 inhibiting monoclonal antibodies Eculizumab and Ravulizumab. However, the duration and optimal dose of treatment are debated, particularly in view of the high costs of the drug. Even if recent studies showed that restrictive use of eculizumab is feasible, there is a clear need for biomarkers identification and protocols for monitoring and predicting disease activity in aHUS and C3G patients.

In summary, new analytic tools for further defining the disease profile in blood, (patients) cells and kidney biopsies are needed.

ELIGIBILITY:
Aim 1

Inclusion Criteria:

* Male and female patients (children and adults) with C3G diagnosis
* Biobank written informed consent

Aim 2 Inclusion criteria

* Male and female patients (children and adults) with aHUS diagnosis in acute phase (before any treatment), or in remission either untreated or undergoing anti-C5 treatment at standard dosing
* Written informed consent Exclusion criteria
* Stx-associated HUS
* TTP (ADAMTS13<10%)
* Plasma therapy within 2 weeks from blood sampling

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Determination of assay sensitivity and specificity | At day 0
  We estimate that 38 VUS/LPV carrying pedigrees should be enough to demonstrate the sensitivity and specificity of the assay for classifying VUS/LPV.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Noris, PhD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noris M, Galbusera M, Gastoldi S, Macor P, Banterla F, Bresin E, Tripodo C, Bettoni S, Donadelli R, Valoti E, Tedesco F, Amore A, Coppo R, Ruggenenti P, Gotti E, Remuzzi G. Dynamics of complement activation in aHUS and how to monitor eculizumab therapy. Blood. 2014 Sep 11;124(11):1715-26. doi: 10.1182/blood-2014-02-558296. Epub 2014 Jul 18. PMID 25037630
- [Background] Iatropoulos P, Daina E, Curreri M, Piras R, Valoti E, Mele C, Bresin E, Gamba S, Alberti M, Breno M, Perna A, Bettoni S, Sabadini E, Murer L, Vivarelli M, Noris M, Remuzzi G; Registry of Membranoproliferative Glomerulonephritis/C3 Glomerulopathy; Nastasi. Cluster Analysis Identifies Distinct Pathogenetic Patterns in C3 Glomerulopathies/Immune Complex-Mediated Membranoproliferative GN. J Am Soc Nephrol. 2018 Jan;29(1):283-294. doi: 10.1681/ASN.2017030258. Epub 2017 Oct 13. PMID 29030465
- [Background] Donadelli R, Pulieri P, Piras R, Iatropoulos P, Valoti E, Benigni A, Remuzzi G, Noris M. Unraveling the Molecular Mechanisms Underlying Complement Dysregulation by Nephritic Factors in C3G and IC-MPGN. Front Immunol. 2018 Oct 15;9:2329. doi: 10.3389/fimmu.2018.02329. eCollection 2018. PMID 30487789
- [Background] Galbusera M, Noris M, Gastoldi S, Bresin E, Mele C, Breno M, Cuccarolo P, Alberti M, Valoti E, Piras R, Donadelli R, Vivarelli M, Murer L, Pecoraro C, Ferrari E, Perna A, Benigni A, Portalupi V, Remuzzi G. An Ex Vivo Test of Complement Activation on Endothelium for Individualized Eculizumab Therapy in Hemolytic Uremic Syndrome. Am J Kidney Dis. 2019 Jul;74(1):56-72. doi: 10.1053/j.ajkd.2018.11.012. Epub 2019 Mar 7. PMID 30851964
- [Background] Piras R, Breno M, Valoti E, Alberti M, Iatropoulos P, Mele C, Bresin E, Donadelli R, Cuccarolo P, Smith RJH, Benigni A, Remuzzi G, Noris M. CFH and CFHR Copy Number Variations in C3 Glomerulopathy and Immune Complex-Mediated Membranoproliferative Glomerulonephritis. Front Genet. 2021 Jun 11;12:670727. doi: 10.3389/fgene.2021.670727. eCollection 2021. PMID 34211499
- [Background] Aiello S, Gastoldi S, Galbusera M, Ruggenenti P, Portalupi V, Rota S, Rubis N, Liguori L, Conti S, Tironi M, Gamba S, Santarsiero D, Benigni A, Remuzzi G, Noris M. C5a and C5aR1 are key drivers of microvascular platelet aggregation in clinical entities spanning from aHUS to COVID-19. Blood Adv. 2022 Jan 8;6(3):866-881. doi: 10.1182/bloodadvances.2021005246. PMID 34852172
- [Background] Piras R, Valoti E, Alberti M, Bresin E, Mele C, Breno M, Liguori L, Donadelli R, Rigoldi M, Benigni A, Remuzzi G, Noris M. CFH and CFHR structural variants in atypical Hemolytic Uremic Syndrome: Prevalence, genomic characterization and impact on outcome. Front Immunol. 2023 Jan 30;13:1011580. doi: 10.3389/fimmu.2022.1011580. eCollection 2022. PMID 36793547
- [Background] Gastoldi S, Aiello S, Galbusera M, Breno M, Alberti M, Bresin E, Mele C, Piras R, Liguori L, Santarsiero D, Benigni A, Remuzzi G, Noris M. An ex vivo test to investigate genetic factors conferring susceptibility to atypical haemolytic uremic syndrome. Front Immunol. 2023 Feb 9;14:1112257. doi: 10.3389/fimmu.2023.1112257. eCollection 2023. PMID 36845135